CLINICAL TRIAL: NCT02313077
Title: A Phase 1, First-in-Human Study to Evaluate the Safety, Tolerability and Immunogenicity of Heterologous Prime-Boost Regimens Using MVA-BN®-Filo and Ad26.ZEBOV Administered in Different Sequences and Schedules in Healthy Adults
Brief Title: A Safety and Immunogenicity Study of Heterologous Prime-Boost Ebola Vaccine Regimens in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR106478; VAC52150EBL1001 (Other: Crucell Holland BV); 2014-004883-39 (EudraCT Number)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Healthy; Ebola viruses; Ebola Viral Disease (EVD); Filoviruses; monovalent vaccine; Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic (MVA-BN) Filo-vector; Safety; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (5):
- Group 1 (Experimental): Participants will receive MVA-BN-filo/ Ad26.ZEBOV (Day 1 /Day 29) or Placebo (Day 1/Day 29).
  Interventions: Biological: MVA-BN-filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 2 (Experimental): Participants will receive MVA-BN-filo/Ad26.ZEBOV (Day 1 /Day 57) or placebo ( Day 1/Day 57).
  Interventions: Biological: MVA-BN-filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 3 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-filo (Day 1/Day 29) or placebo (Day 1/Day 29).
  Interventions: Biological: MVA-BN-filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 4 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-filo (Day 1/Day 57) or placebo (Day 1/Day 57).
  Interventions: Biological: MVA-BN-filo; Biological: Ad26. ZEBOV; Other: Placebo
- Group 5 (Experimental): Participants will receive Ad26.ZEBOV/ MVA-BN-filo (Day 1/Day 15).
  Interventions: Biological: MVA-BN-filo; Biological: Ad26. ZEBOV

INTERVENTIONS:
Biological: MVA-BN-filo — One 0.5 mL intramuscular (IM) injection of 1E8 (50%Tissue Culture Infectious Dose [TCID50]) on Day 1 (Groups 1 and 2), or on Day 29 (Group 3), or on Day 57 (Group 4), or on Day 15 (Group 5).
Biological: Ad26. ZEBOV — One 0.5 mL IM injection of 5E10 viral particles (vp) on Day 1 (Groups 3, 4 and 5), or on Day 29 (Group 1), or on Day 57 (Group 2).
Other: Placebo — One 0.5 mL IM injection of 0.9% saline on Day 1 and 29 (Groups 1 and 3), or on Day 1 and 57 (Groups 2 and 4).
  Arms: Group 1; Group 2; Group 3; Group 4

SUMMARY:
The purpose of this study is to test the safety and immunogenicity of MVA-BN-Filo and Ad26.ZEBOV as heterologous prime-boost vaccine regimens in healthy adult participants.

DETAILED DESCRIPTION:
This first-in-human study consists of 2 parts: 1) The main study, which is randomized, placebo-controlled, observer-blind; 2) A sub-study, which is open-label, uncontrolled, non-randomized study evaluating the safety, tolerability, and immunogenicity of MVA-BN-Filo and Ad26.ZEBOV administered in different sequences and schedules to healthy adult participants. The study consists of a Screening period (up to 28 days in the main study and up to 56 days in the sub-study), a vaccination period in which participants will be vaccinated at baseline (Day 1) followed by a boost on Day 15, 29 or 57, and a post-boost follow-up until all participants have had their 21-day post-boost visit (Day 36, 50 or Day 78). The total duration of the study will be about 1 year for participants who received vaccine and about 3 months for participants who received placebo. Safety will be monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy on the basis of physical examination, medical history, and the investigator's clinical judgment
* Women of childbearing potential must have a negative serum β-human chorionic gonadotropin pregnancy test at screening, a negative urine pregnancy test immediately prior to each study vaccine administration, and practice adequate birth control measures from 28 days before the prime vaccination until at least 3 months after the boost vaccination as specified in the study protocol. If not heterosexually active at screening, must agree to practice adequate birth control measures if they become heterosexually active during their participation in the study (from screening onwards until at least 3 months after the boost vaccination). Agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction from screening onwards until at least 3 months after the boost vaccination
* Women of non-childbearing potential, defined as postmenopausal (>45 years of age with amenorrhea for ≥2 years or any age with amenorrhea for ≥6 months and serum follicle-stimulating hormone [FSH] >40 mIU/mL) or surgically sterile (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), are not required to use the birth control methods as specified in the study protocol
* A man who is sexually active with a woman of childbearing potential and who has not had a vasectomy must agree to use a double-barrier method of birth control, such as either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository. In case the female partner is using an adequate method of birth control, a single-barrier method of birth control for the male subject is acceptable. Men must also agree not to donate sperm from screening onwards until at least 3 months after the boost vaccination
* Must be available and willing to participate for the duration of the study visits and follow-up, provide verifiable identification, and have a means to be contacted

Exclusion Criteria:

* Has been vaccinated with a candidate Ebola vaccine
* Has been diagnosed with Ebola disease or exposed to Ebola including travel to West Africa in the last 12 months. West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, and Sierra Leone
* Has received any Ad26- or MVA-based candidate vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines), including known allergy to egg or aminoglycosides
* A woman who is pregnant or breast-feeding, or planning to become pregnant while enrolled in the study or within 3 months after the boost vaccination
* History of diabetes mellitus type 1 or type 2, including cases controlled with diet alone; thyroidectomy, or thyroid disease requiring medication during the last 12 months; uncontrolled hypertension as defined in the study protocol; or, major psychiatric illness and/or substance abuse problems during the past 12 months that in the opinion of the investigator would preclude participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2015-04-17 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 21 days after the 2nd vaccination (Day 36 for Group 5 or Day 50 for Groups 1 and 3 or Day 78 for Groups 2 and 4)
Number of participants with serious adverse events | Up to the end of long-term follow-up (Day 360)
Number of participants with reactogenicity (ie, solicited local and systemic adverse events) | Up to 1 week after each study vaccine administration

SECONDARY OUTCOMES:
Immune responses to the study vaccine regimens as measured by a virus neutralization assay | Groups 1 and 3:Day 1(pre-vaccination), 8, 29(pre-vaccination), 36, 50, 180, 240, 360; Groups 2 and 4:Day 1(pre-vaccination), 8, 29, 57(pre-vaccination), 64, 78, 180, 240, 360; Group 5:Day 1(pre-vaccination), 8, 15(pre-vaccination), 22, 36, 180, 240, 360
Immune responses to the study vaccine regimens measured by an enzyme-linked immunosorbent assay (ELISA) | Groups 1 and 3:Day 1(pre-vaccination), 8, 29(pre-vaccination), 36, 50, 180, 240, 360; Groups 2 and 4:Day 1(pre-vaccination), 8, 29, 57(pre-vaccination), 64, 78, 180, 240, 360; Group 5:Day 1(pre-vaccination), 8, 15(pre-vaccination), 22, 36, 180, 240, 360
Immune responses to the study vaccine regimens as measured by an enzyme-linked immunospot (ELISpot) assay | Groups 1 and 3:Day 1(pre-vaccination), 8, 29(pre-vaccination), 36, 50, 180, 240, 360; Groups 2 and 4:Day 1(pre-vaccination), 8, 29, 57(pre-vaccination), 64, 78, 180, 240, 360; Group 5:Day 1(pre-vaccination), 8, 15(pre-vaccination), 22, 36, 180, 240, 360

CONTACTS AND LOCATIONS:
Overall Officials: Crucell Holland BV Clinical Trial, Study Director — Crucell Holland BV
Locations (1):
- Oxford, United Kingdom

REFERENCES:
- [Derived] Wagstaffe HR, Clutterbuck EA, Bockstal V, Stoop JN, Luhn K, Douoguih M, Shukarev G, Snape MD, Pollard AJ, Riley EM, Goodier MR. Ebola virus glycoprotein stimulates IL-18-dependent natural killer cell responses. J Clin Invest. 2020 Jul 1;130(7):3936-3946. doi: 10.1172/JCI132438. PMID 32315287
- [Derived] Milligan ID, Gibani MM, Sewell R, Clutterbuck EA, Campbell D, Plested E, Nuthall E, Voysey M, Silva-Reyes L, McElrath MJ, De Rosa SC, Frahm N, Cohen KW, Shukarev G, Orzabal N, van Duijnhoven W, Truyers C, Bachmayer N, Splinter D, Samy N, Pau MG, Schuitemaker H, Luhn K, Callendret B, Van Hoof J, Douoguih M, Ewer K, Angus B, Pollard AJ, Snape MD. Safety and Immunogenicity of Novel Adenovirus Type 26- and Modified Vaccinia Ankara-Vectored Ebola Vaccines: A Randomized Clinical Trial. JAMA. 2016 Apr 19;315(15):1610-23. doi: 10.1001/jama.2016.4218. PMID 27092831